CLINICAL TRIAL: NCT06297252
Title: Prevalence of Psychiatric Disorders During Pregnancy at 2nd Trimester Ultrasound: a Feasibility Study in the General Population
Acronym: GROUP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Beziers Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL23_0189
Record Dates: First submitted 2024-02-19; First posted 2024-03-07 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy
Keywords: Mental Disorders During Pregnancy; perinatology; Social Vulnerability; Mental Disorders; pregnancy
MeSH Terms: conditions — Mental Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant adults (Experimental): Adults women with an ongoing pregnancy who are scheduled for a T2 ultrasound, regardless of known history or pregnancy context (normal or pathological).
  Interventions: Diagnostic Test: standardized clinical psychiatric evaluations; Diagnostic Test: self-administered psychiatric questionnaire assessments; Other: blood sampling

INTERVENTIONS:
Diagnostic Test: standardized clinical psychiatric evaluations — The intervention consists of a psychiatric consultation including :
  * assessment of psychiatric disorders using a MINI test
  * information gathering (medical, obstetrical and family history, expected term of pregnancy).
  * assessment of suicidal behaviour using the Columbia-Suicide Severity Rating Scale (CSSR-S)
  * collection of negative life events over the past 12 months, assessed using the Paykel questionnaire
Diagnostic Test: self-administered psychiatric questionnaire assessments — * EPICES Score: (Evaluation de la Précarité et des Inégalités de santé dans les Centres d'Examens de Santé):
  * MIBS: (Mother to Infant Bonding Scale)
  * PAI: (Prenatal Attachment Inventory)
  * EDEQ: (Eating Disorder Examination Questionnaire)
  * PCL-5: (Post-traumatic Stress Disorder Checklist for DSM-V)
  * MARS: (Medication Adherence Rating Scale)
  * EPDS: (Edinburgh Postnatal Depression Scale)
Other: blood sampling — A blood sample is taken to form an optional biological collection, comprising 3 samples:
  * A tube to collect RNA from whole blood.
  * A tube to collect serum
  * A tube to collect native DNA

SUMMARY:
Young women represent a population at risk of psychiatric disorders, the first signs of which often appear between the ages of 15 and 25. Psychiatric disorders are a major source of disability and healthcare costs.

The perinatal period is an additional period of psychological vulnerability, during which women are at increased risk of developing or worsening psychiatric disorders. Unfortunately, psychiatric disorders seem to be largely under-diagnosed during this period, and therefore under-treated.

The goal of this Prospective multicenter study is to determine the prevalence of the presence of at least one characterized psychiatric disorder, as defined by the use of the Mini International Neuropsychiatric Interview (MINI), in remission or not, during pregnancy, at the time of the second-trimester ultrasound (T2 ultrasound) based on a standardized clinical assessment.

Participants will complete self-questionnaires and have a standardized psychiatric evaluation at T2 ultrasound and at 2 months postpartum.

DETAILED DESCRIPTION:
Young women represent a population at risk of psychiatric disorders, the first signs of which often appear between the ages of 15 and 25. Psychiatric disorders are a major source of disability and healthcare costs. They are often comorbid, and can be complicated by suicidal behaviour. Delays in diagnosis are common, significantly worsening the prognosis and increasing the societal cost of these disorders.

The perinatal period is an additional period of psychological vulnerability, during which women are at increased risk of developing or worsening psychiatric disorders. Unfortunately, these disorders seem to be largely under-diagnosed during this period, and therefore under-treated.

To date, psychiatric diagnoses are exclusively clinical. They can be facilitated by screening questionnaires, the sensitivity and specificity of which are highly heterogeneous and sometimes poorly understood in the perinatal period and in the general population of pregnant women. What's more, several studies have shown that clinical diagnosis in everyday practice often lacks sensitivity when compared with standardized assessments, i.e. those based on a structured and reproducible diagnostic approach, which is longer and more costly, such as the MINI (Mini International Neuropsychiatric Interview).

The state of knowledge on the epidemiology of psychiatric disorders in the perinatal period suffers from many imperfections. The vast majority of studies focus exclusively on postpartum depression. This project, on the other hand, focuses on the diagnosis of any psychiatric disorder characterized by a standardized diagnostic interview (validated and reproducible, like the MINI) carried out by a professional trained in the clinical management of psychiatric disorders.

Biomarkers, in particular to aid differential diagnosis, are being developed and are a source of hope for improving the quality of screening; but the results are rarely replicated in independent cohorts or from biological banks associated with quality clinical data.

Our hypothesis is that the prevalence of psychiatric disorders (current or in remission), in this population, is at least 20% and that more than half of these disorders are unknown.

From a practical point of view, it aims to improve assessments of psychiatric vulnerabilities within the two main public maternity hospitals in the Hérault department in France.

From a scientific point of view, it will provide an opportunity to create a highly original bank of biological samples, opening up interesting research prospects in psychiatry, but also well beyond, given the specific nature of the population concerned.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 years and over
* Pregnant and consulting for scheduled second trimester ultrasound
* Able to read and write with a good knowledge of French

Exclusion Criteria:

* Unable to understand French
* Illiterate
* Underage patient at time of second trimester ultrasound
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient not affiliated to or not benefiting from a social security scheme
* Refusal of consent after information
* Participant in another research project with an ongoing exclusion period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women only
Enrollment: 140 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-10-24 (Estimated)

PRIMARY OUTCOMES:
To determine the prevalence of the presence of at least one characterized psychiatric disorder, in remission or not, during pregnancy, at the time of the second-trimester ultrasound (T2 ultrasound) based on a standardized clinical assessment. | Baseline (T2 ultrasound)
  Presence of at least one psychiatric disorder (evaluated by the MINI), of any kind, in remission or not, during pregnancy, at the time of the T2 ultrasound.
  The MINI score verifies the presence or absence of criteria for the most common psychiatric illnesses and assess the 17 most common psychiatric disorders and suicidality in DSM-III-R, DSM-IV and DSM-5 and ICD-10.
  * Affective Disorders, Psychotic
  * Agoraphobia
  * Alcoholism
  * Anorexia Nervosa
  * Antisocial Personality Disorder
  * Anxiety Disorders
  * Bipolar and Related Disorders
  * Bipolar Disorder
  * Bulimia Nervosa
  * Depressive Disorder, Major
  * Mania
  * Obsessive-Compulsive Disorder
  * Panic Disorder
  * Phobia, Social
  * Psychotic Disorders
  * Self-Injurious Behavior
  * Stress Disorders, Post-Traumatic
  * Substance-Related Disorders
  * Suicidal Ideation

SECONDARY OUTCOMES:
To determine the prevalence of each psychiatric disorder characterized during pregnancy at the time of the second-trimester ultrasound, based on a standardized clinical assessment. | Baseline (T2 ultrasound)
  Standardized clinical assessment includes MINI, Columbia-Suicide Severity Rating Scale (CSSR-S) questionnaire used for suicide assessment (scale from 0 to 5 (highest suicidal risk)), Negative life events in the last 12 months will be assessed using the Paykel questionnaire, and a medical examination by a psychiatrist.
  All these elements are used together to diagnose psychiatric disorders and determine their individual prevalence.
  The MINI score verifies the presence or absence of criteria which assess the 17 most common psychiatric disorders and suicidality : Affective Disorders, Psychotic, Agoraphobia, Alcoholism, Anorexia Nervosa, Antisocial Personality Disorder, Anxiety Disorders, Bipolar and Related Disorders, Bipolar Disorder, Bulimia Nervosa, Depressive Disorder, Major, Mania, Obsessive-Compulsive Disorder, Panic Disorder, Phobia Social, Psychotic Disorders, Self-Injurious Behavior, Stress Disorders, Post-Traumatic, Substance-Related Disorders, Suicidal Ideation
Determine comorbidity profiles across all pathologies, describing whether there are patient groups based on these profiles. | Baseline (T2 ultrasound) and 2 months postpartum
  Clustering methods (unsupervised classification) will be used to construct homogeneous subgroups of subjects according to comorbidities.
Compare the prevalence of psychiatric disorders unknown to the obstetrics team with the prevalence of known psychiatric disorders in pregnant patients at the time of T2 ultrasound. | Baseline (T2 ultrasound)
  Prevalence of diagnoses unknown to the obstetrical team and/or not documented in the obstetrical record.
Compare the prevalence of psychiatric disorders unknown to the patient with the prevalence of known psychiatric disorders in pregnant patients at the time of T2 ultrasound. | Baseline (T2 ultrasound)
  Prevalence of diagnoses unknown to the patient.
Compare the prevalence of psychiatric disorders unknown to the general practitioner with the prevalence of known psychiatric disorders in pregnant patients at the time of T2 ultrasound. | Baseline (T2 ultrasound)
  Prevalence of diagnoses unknown to the general practitioner
Assess patients' medication compliance using self-administered questionnaires (MARS). | Baseline (T2 ultrasound) and 2 months post partum
  Medication Adherence Report Scale (MARS) 10 items questionnaire with scores ranging from 0 (lowest adhesion) to 10 (highest)
Assess patients' treatment beliefs using self-administered questionnaires (BMQ). | Baseline (T2 ultrasound) and 2 months post partum
  Belief on Medicine Questionnaire (BMQ) with 18 items, with a scores ranging from 18 (lowest belief) to 90 (highest)
Determine the sociodemographic, psychological, psychiatric, medical and obstetric factors, as well as those associated with access to care and the care pathway associated with known or unknown diagnoses during pregnancy. | Baseline (T2 ultrasound) and 2 months post partum
  Evaluation of socio-demographic dimension with the French score : Evaluation of precariousness and health inequalities in health examination centers (Evaluation de la Précarité et des Inégalités de santé dans les Centres d'Examens de Santé EPICES). This score assesses the marital status, place of residence, level of education, current employment situation, social security coverage, factors of precariousness.
Determine the properties (sensitivity) of screening questionnaires (EPDS) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the sensitivity value will be calculated along with the associated 95% confidence intervals.
  - Accuracy of the Edinburgh Postnatal Depression Scale (EPDS) is a 10 items questionnaire with scores ranging from 0 (lowest depression score) to 30 (Highest)
Determine the properties (specificity) of screening questionnaires (EPDS) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the specificity value will be calculated along with their associated 95% confidence intervals.
  - Accuracy of the Edinburgh Postnatal Depression Scale (EPDS) is a 10 items questionnaire with scores ranging from 0 (lowest depression score) to 30 (Highest)
Determine the properties (positive predictive value) of screening questionnaires (EPDS) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the positive predictive value will be calculated along with their associated 95% confidence intervals.
  - Accuracy of the Edinburgh Postnatal Depression Scale (EPDS) is a 10 items questionnaire with scores ranging from 0 (lowest depression score) to 30 (Highest)
Determine the properties (negative predictive value) of screening questionnaires (EPDS) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains negative predictive value will be calculated along with their associated 95% confidence intervals.
  - Accuracy of the Edinburgh Postnatal Depression Scale (EPDS) is a 10 items questionnaire with scores ranging from 0 (lowest depression score) to 30 (Highest)
Determine the properties (sensitivity) of screening questionnaires ( MDQ) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the sensitivity will be calculated along with their associated 95% confidence intervals.
  - Mood Disorder Questionnaire (MDQ) composed of 15-items with scores ranging from 0 (lowest risk of mood disorder) to 13 (Highest)
Determine the properties (specificity) of screening questionnaires ( MDQ) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the specificity will be calculated along with their associated 95% confidence intervals.
  - Mood Disorder Questionnaire (MDQ) composed of 15-items with scores ranging from 0 (lowest risk of mood disorder) to 13 (Highest)
Determine the properties (positive predictive value) of screening questionnaires ( MDQ) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the positive predictive value will be calculated along with their associated 95% confidence intervals.
  - Mood Disorder Questionnaire (MDQ) composed of 15-items with scores ranging from 0 (lowest risk of mood disorder) to 13 (Highest)
Determine the properties (negative predictive value) of screening questionnaires ( MDQ) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the negative predictive value will be calculated along with their associated 95% confidence intervals.
  - Mood Disorder Questionnaire (MDQ) composed of 15-items with scores ranging from 0 (lowest risk of mood disorder) to 13 (Highest)
Determine the properties (sensitivity) of screening questionnaires (PCL-5) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the sensitivity will be calculated along with their associated 95% confidence intervals.
  - Post-traumatic Stress Disorder Checklist for DSM-V (PCL-5) is a 20 items questionnaires with scores ranging from 0 (lowest risk of PTSD) to 80 (Highest)
Determine the properties (specificity) of screening questionnaires (PCL-5) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the specificity will be calculated along with their associated 95% confidence intervals.
  - Post-traumatic Stress Disorder Checklist for DSM-V (PCL-5) is a 20 items questionnaires with scores ranging from 0 (lowest risk of PTSD) to 80 (Highest)
Determine the properties (positive predictive value) of screening questionnaires (PCL-5) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the positive predictive value will be calculated along with their associated 95% confidence intervals.
  - Post-traumatic Stress Disorder Checklist for DSM-V (PCL-5) is a 20 items questionnaires with scores ranging from 0 (lowest risk of PTSD) to 80 (Highest)
Determine the properties (negative predictive value) of screening questionnaires (PCL-5) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the negative predictive value will be calculated along with their associated 95% confidence intervals.
  - Post-traumatic Stress Disorder Checklist for DSM-V (PCL-5) is a 20 items questionnaires with scores ranging from 0 (lowest risk of PTSD) to 80 (Highest)
Determine the properties (sensitivity) of screening questionnaires (EDEQ) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the sensitivity will be calculated along with their associated 95% confidence intervals.
  - Eating Disorder Examination Questionnaire (EDE-Q) is a 28 items questionnaires with a higher score indicating more problematic eating difficulties.
Determine the properties (specificity) of screening questionnaires (EDEQ) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, specificity will be calculated along with their associated 95% confidence intervals.
  - Eating Disorder Examination Questionnaire (EDE-Q) is a 28 items questionnaires with a higher score indicating more problematic eating difficulties.
Determine the properties (positive predictive value) of screening questionnaires (EDEQ) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the positive predictive value will be calculated along with their associated 95% confidence intervals.
  - Eating Disorder Examination Questionnaire (EDE-Q) is a 28 items questionnaires with a higher score indicating more problematic eating difficulties.
Determine the properties (negative predictive value) of screening questionnaires (EDEQ) for psychiatric disorders in this population. | Baseline (T2 ultrasound) and 2 months post partum
  the results of these tests according to the thresholds already established in the literature will be compared with the results of the corresponding MINI sub-domains, and the negative predictive value will be calculated along with their associated 95% confidence intervals.
  - Eating Disorder Examination Questionnaire (EDE-Q) is a 28 items questionnaires with a higher score indicating more problematic eating difficulties.
Compare mother-child bonding difficulties between patients with and without a psychiatric diagnosis at the time of the study, using scales (PAI). | 2 months post partum
  - Personality Assessment Inventory (PAI) 21 items questionnaire with scores ranging from 21 (the least feeling for their baby) to 84 (Highest)
Compare mother-child bonding difficulties between patients with and without a psychiatric diagnosis at the time of the study, using scales (MIBS). | 2 months post partum
  - Mother-to-Infant Bonding Scale (MIBS) 8 items questionnaire with scores ranging from 0 (highest Bonding) to 24 (Lowest)
Describe how the study will be carried out, either in person or by teleconsultation, and the reasons for this choice. | Baseline (T2 ultrasound) and 2 months post partum
  Percentage of face-to-face and teleconsultation consultations and the reasons for this choice
Determine the prevalence of each psychiatric disorder at two months post-inclusion based on a standardized clinical assessment. | 2 months post partum
  Standardized clinical assessment includes MINI, Columbia-Suicide Severity Rating Scale (CSSR-S) questionnaire used for suicide assessment (scale from 0 to 5 (highest suicidal risk)), Negative life events in the last 12 months will be assessed using the Paykel questionnaire, and a medical examination by a psychiatrist.
  All these elements are used together to diagnose psychiatric disorders and determine their individual prevalence.
  The MINI score verifies the presence or absence of criteria which assess the 17 most common psychiatric disorders and suicidality : Affective Disorders, Psychotic, Agoraphobia, Alcoholism, Anorexia Nervosa, Antisocial Personality Disorder, Anxiety Disorders, Bipolar and Related Disorders, Bipolar Disorder, Bulimia Nervosa, Depressive Disorder, Major, Mania, Obsessive-Compulsive Disorder, Panic Disorder, Phobia Social, Psychotic Disorders, Self-Injurious Behavior, Stress Disorders, Post-Traumatic, Substance-Related Disorders, Suicidal Ideation

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Belzeaux, MD PhD, Study Director — University Hospital, Montpellier
Locations (2):
- France (2):
  - Centre Hospitalier de Béziers, Béziers
  - University Hospital of Montpellier, Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knabe L, Tanaka C, Tebeka S, Neilson S, Cauvin C, Mercier N, Cayron D, Savelli M, Deruelle P, Fuchs F, Pissarra J, Molinari N, Belzeaux R. Prevalence of psychiatric disorders during pregnancy-a feasibility study at second trimester ultrasound in the general population (GROUP study): study protocol. BMJ Open. 2025 Feb 20;15(2):e091923. doi: 10.1136/bmjopen-2024-091923. PMID 39979054